CLINICAL TRIAL: NCT03185611
Title: Effectiveness of Rifaximin Combined With Thiopurine on Preventing Postoperative Endoscopic Recurrence in Crohn's Disease Patients With Risk Factor for Recurrence: A Multicenter Randomized Controlled Trial
Brief Title: Effectiveness of Rifaximin Combined With Thiopurine on Preventing Postoperative Recurrence in Crohn's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Peking Union Medical College Hospital (Other); Xijing Hospital (Other); Shanghai 10th People's Hospital (Other); RenJi Hospital (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-ZSLY-06
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Rifaximin; Azathioprine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin and Thiopurine (Experimental): Prescribed Rifaximin (600mg, twice daily) combined with Azathioprine (2.0-2.5mg/kg/day) for 3 months after surgery, and then Azathioprine monotherapy (2.0-2.5mg/kg/day) for the next 3months.
  Interventions: Drug: Rifaximin; Drug: Azathioprine
- Thiopurine (Active Comparator): Prescribed Azathioprine (2.0-2.5mg/kg/day) for 6 months after surgery.
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Rifaximin — Antibiotics
  Arms: Rifaximin and Thiopurine
Drug: Azathioprine — immunomodulator

SUMMARY:
Some studies have shown that rifaximin is effective in the management of Crohn's Disease. Meanwhile, its adverse effect is tolerable. But no study has been conducted to assess its effect on preventing postoperative recurrence. Thus, we conduct a randomised controlled study to assess the effect of rifaximin combined with thiopurine on preventing postoperative endoscopic recurrence in Crohn's disease, compared with thiopurine. The primary endpoint is the rate of endoscopic recurrence at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with Crohn's disease undergoing intestinal resection of all macroscopic diseased bowel, with an endoscopically accessible ileocolic anastomosis;
2. Enrolled patients must have one or more risk factor for the development of postoperative recurrence including penetrating disease behaviour, prior bowel resection, and active smoking.

Exclusion Criteria:

1. Severe comorbidities;
2. With a stoma;
3. With malignancy;
4. Pregnancy;
5. Intolerant of thiopurine drugs;
6. With contraindication of using rifaximin or thiopurine drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
difference of incidence of endoscopic recurrence | 6 months after surgery
  Endoscopic recurrence was defined by a score ≥i2 according to endoscopic recurrence score developed by Rutgeerts et al.

SECONDARY OUTCOMES:
Adverse effect | 6 months after surgery
  Adverse effect of Rifaximin

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guanzhou, Guangdong, China